CLINICAL TRIAL: NCT04984915
Title: The Long-term Prognostic Value of CaIMR in Patients With ST-segment Elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention
Brief Title: The Usefulness of CaIMR in Patients With STEMI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhibing Lu, The chief of cardiology department, Zhongnan Hospital
Other Study IDs: 2021075
Record Dates: First submitted 2021-06-06; First posted 2021-08-02 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: CaIMR; Prognosis; ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The coronary artery system is composed of three different types of blood vessels, namely epicardial arteries, arterioles and capillaries. Compared with epicardial arteries, arterioles and capillaries are lower than the resolution of current angiography systems, so angiography cannot be used for visualization. Existing studies have shown that coronary microcirculation plays an extremely important role in maintaining full myocardial perfusion. Coronary microvascular disorders can lead to myocardial hypoperfusion and ischemia, and are related to the poor prognosis of patients with coronary heart disease. At present, there is no technology that can directly detect the state of the coronary microcirculation in the human body, but the coronary microcirculation function can be indirectly assessed through two invasive and non-invasive methods. Among them, the index of microcirculation resistance (IMR) is widely used to evaluate coronary microcirculation function [3]. However, in the case of epicardial stenosis, accurate determination of IMR requires knowledge of coronary artery contraction pressure (Pw). However, measuring IMR is an invasive examination technique, and measuring IMR requires high technical requirements for the operator. Therefore, the CaIMR value obtained by AI technology can well overcome this limitation, and the existing data show that the CaIMR value has a good correlation with the IMR value. However, CaIMR has a clinical prognosis for patients with acute ST-segment elevation myocardial infarction. The predictive value of CaIMR has not yet been explored. This project aims to evaluate the application value of CaIMR in predicting the occurrence of adverse cardiovascular events in patients with acute ST-segment elevation myocardial infarction after percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are clinically diagnosed with acute ST-segment elevation myocardial infarction and are planned to undergo PCI;
* Volunteer to participate and sign the informed consent

Exclusion Criteria:

* Coronary angiography suggests that it is not suitable for PCI;
* Have performed CABG surgery in the past;
* Lesion of left or right coronary ostium;
* The target vessel is an infarct-related artery (old or acute myocardial infarction recovery period);
* The immediate effect of target vessel PCI is not ideal (such as: final TIMI blood flow <grade 3, dissection with restricted blood flow, side branch occlusion with diameter> 1.5 mm, distal embolism or thrombus shown by angiography);
* Severe systemic infection;
* Patients with malignant wasting disease whose estimated survival time is less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the inclusion and exclusion criteria are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The composite endpoint of all-cause death and heart failure rehospitalization | 1 year after surgery
  The composite endpoint of all-cause death and heart failure rehospitalization

SECONDARY OUTCOMES:
The composite endpoint of all-cause death and heart failure rehospitalization | 1 month after surgery
  The composite endpoint of all-cause death and heart failure rehospitalization
All-cause death | 1 year after surgery
  All-cause death
All-cause death | 1 month after surgery
  All-cause death
Heart failure rehospitalization | 1 year after surgery
  Heart failure rehospitalization
Heart failure rehospitalization | 1 month after surgery
  Heart failure rehospitalization
Cardiogenic Rehospitalization | 1 year after surgery
  Cardiogenic Rehospitalization
Cardiogenic Rehospitalization | 1 month after surgery
  Cardiogenic Rehospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China